CLINICAL TRIAL: NCT04262128
Title: Prolonged Sedentary Behavior in Older Women With and Without Type 2 Diabetes: Knowledge, Engagement, and Relationship to Cardiometabolic Risk
Brief Title: Sedentary Behavior in Older Women With and Without Type 2 Diabetes
Acronym: SitWise
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 19-2758
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus, Type 2; Healthy
Keywords: diabetes; sedentary behavior; cardiovascular disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Sedentary Behavior; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Type 2 Diabetes Mellitus: women age 60-75 years with uncomplicated type 2 diabetes mellitus
- Healthy Controls: healthy women age 60-75 years

SUMMARY:
Sedentary behavior has been linked to cardiovascular morbidity and mortality, and is particularly common in older adults with type 2 diabetes. The purpose of this observational, mixed-methods study is to better understand the relationship between prolonged sedentary behavior and cardiovascular and metabolic health in older women.

DETAILED DESCRIPTION:
The investigators will recruit 20 women age 60-75 years, n=10 with uncomplicated type 2 diabetes (T2D) and n=10 healthy controls. Participants will wear two accelerometers and a continuous glucose monitor (CGM) for two different periods of 7 days for objective assessment of physical activity, sedentary behavior, and blood glucose, respectively, and complete a graded exercise test (cardiorespiratory fitness), assessment of insulin sensitivity (hyperinsulinemic-euglycemic clamp) and single leg exercise using near-infrared spectroscopy (microvascular function). Participants will also complete a semi-structured qualitative interview to understand knowledge and attitudes toward sedentary behavior and questionnaires to assess the relationship between modifiable psychological and behavioral factors and sedentary behavior.

The aims of the study are to:

1. Compare objectively-measured, free-living physical activity and sedentary behavior between older women with and without T2D.
2. Evaluate the relationship between prolonged bouts of sedentary behavior, cardiorespiratory fitness, glucose control, insulin sensitivity, and skeletal muscle microvascular function in older women with and without T2D.
3. Assess knowledge and attitudes toward sedentary behavior and characterize the relationship between knowledge and attitudes toward sedentary behavior and modifiable psychological and behavioral factors in older women with T2D.
4. Evaluate the relationship between sedentary behavior, mood states, and meaning salience during "normal" life and the period of confinement imposed by the COVID-19 epidemic.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 60-75 years
* Postmenopausal (self-reported)
* BMI between 25-40 kg/m2
* Participants with T2D:
* T2D confirmed via chart review
* T2D diet controlled or treated with the following acceptable medication treatments: metformin, sulfonylureas, glinides, or glucose absorption blockers

Exclusion Criteria:

* Male
* Age <60 or >75 years
* Type 1 diabetes
* Control participants only - HbA1C ≥ 5.7%
* Use of beta blockers or centrally-acting calcium channel blockers (i.e., diltiazem, verapamil) due to potential blunting of cardiorespiratory fitness assessments
* Use of hormone replacement therapy (e.g., estrogen, progesterone, testosterone) (within the past 5 years)
* Taking insulin, thiazolidinediones (e.g., rosiglitazone), glucagon-like peptide-1 (GLP1) agonists (e.g., exenatide), dipeptidyl peptidase-4 (DPP4) inhibitors (e.g., sitagliptin) or any medication for the treatment of T2D other than those listed above in the inclusion criteria
* Uncontrolled hypertension at rest (systolic >160 or diastolic >110 mmHg)
* Obstructive pulmonary disease or asthma with a forced expiratory volume in 1 second (FEV1)/forced vital capacity (FVC) ratio <70% of predicted
* Any of the following conditions:
* Uncontrolled T2D (HbA1C >9.0%)
* Unstable angina
* Recent myocardial infarction, cardiac surgery, or vascular surgery (<3 months)
* Heart failure
* Peripheral artery disease (based on report of symptomatic claudication or ankle brachial index testing)
* Anemia (tHb <10 mg/dL)
* Hepatic or renal disease
* Severe arthritis or mobility impairment that would interfere with exercise testing
* Current tobacco or marijuana use or nicotine use within the last year
* Dementia or evidence of cognitive impairment (Mini-Cog score < 3)
* Engaging in >150 minutes/week of moderate to vigorous physical activity (assessed via Low-Level Physical Activity Recall questionnaire)

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy women and women with T2D age 60-75 years.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
time sedentary measured via triaxial accelerometer | 7 days
average sedentary bout length measured via triaxial accelerometer | 7 days
cardiorespiratory fitness | 8-12 minutes
  peak volume of oxygen consumption (VO2 peak) in ml/kg/min measured via graded exercise test
insulin sensitivity | 3 hours
  glucose infusion rate in mg/kg/min as measured via hyperinsulinemic-euglycemic clamp
change in skeletal muscle deoxygenated hemoglobin concentration during single leg calf exercise measured via near-infrared spectroscopy | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Mary O Whipple, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No